CLINICAL TRIAL: NCT04017247
Title: A Comparison Between Continuous Versus Intermittent Oxytocin Infusion for Induction of Labor
Brief Title: Continuous Versus Intermittent Oxytocin Infusion for Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0308-19-RMB
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Induced; Birth
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent treatment (Active Comparator): Infusion of oxytocin for 6 hours at a time until patient delivers.
  Interventions: Drug: Oxytocin
- Continous treatment (Active Comparator): Infusion of oxytocin continuously from patient admission for 16 hours.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intermittent oxytocin Infusion
  Arms: Intermittent treatment
Drug: Oxytocin — Continous oxytocin Infusion for 16 hours
  Arms: Continous treatment

SUMMARY:
The study will compare 2 treatment modalities. One group will receive the routine protocol of intermittent pitocin induction for 6 hours and the second group will receive continous pitocin infusion for 16 hours.

The primary aim is to observe which protocol leads to the fastest delivery and evaluate the time in each group from induction to delivery.

DETAILED DESCRIPTION:
After singing an informed consent, and prior to IOL initiation, study participants were randomly assigned (1:1) to receive either intermittent or continuous Oxytocin infusion. Both groups received the same primary infusion dose of Oxytocin 1.0 with an incremental increase of 2.5 every 30 minutes until 20, titered to a target of 3-5 contractions in a 10 minute period. During Oxytocin infusion, fetal heart rate was continuously monitored. Artificial ROM was performed according to the accepted indications, local protocol and by the staff physician discretion who was in charge on the labor ward at that time, regardless of oxytocin initiation time. In the intermittent Oxytocin infusion group, Oxytocin was discontinued after 8 h if the patient did not go into active labor during by that time, and renewed 4 h later. In the continuous infusion group, patients received a continuous Oxytocin infusion for 16 h. If they did not go into active labor within this frame time, Oxytocin was discontinued for 4 hours and then resumed. In addition, during Oxytocin infusion, sodium levels were monitored every 8 h.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton pregnancy that are admitted for induction or augmentation of labor.
2. Women at gestational age 370/7 or more.
3. Vertex presentation.

Exclusion Criteria:

1. Age under 18 or over 45.
2. High order gestation.
3. Women with contraindication for vaginal delivery.
4. Active labor.
5. Women with a uterine scar.
6. Multiparity(> 5 deliveries).
7. Documented fetal anomalies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 153 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Delivery within 24 hours | from admission up to 24 hours postpartum
  The percentage of women delivering within 24 hours.

SECONDARY OUTCOMES:
latent phase of labor. | from admission up to 24 hours postpartum
  Length of latent phase of labor.
active phase of labor. | from admission up to 24 hours postpartum
  Length of active phase of labor.
caesarian deliveries | from admission up to 24 hours postpartum
  The rate of caesarian deliveries.
instrumental deliveries | from admission up to 24 hours postpartum
  The rate of instrumental deliveries.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Principal Investigator
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bachar G, Abu-Rass H, Farago N, Justman N, Buchnik G, Chen YS, David CB, Goldfarb N, Khatib N, Ginsberg Y, Zipori Y, Weiner Z, Vitner D. Continuous vs intermittent induction of labor with oxytocin in nulliparous patients: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Dec;5(12):101176. doi: 10.1016/j.ajogmf.2023.101176. Epub 2023 Oct 7. PMID 37813304